CLINICAL TRIAL: NCT05128825
Title: A Phase 2 Open-Label, Multicenter Study To Evaluate Efficacy And Safety Of ZN-c3 In Subjects With High-Grade Serous Ovarian, Fallopian Tube, Or Primary Peritoneal Cancer (DENALI / ZN-c3-005 / GOG-3066)
Brief Title: A Study of Azenosertib (ZN-c3) in Subjects With Platinum-Resistant High-Grade Serous Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Acronym: DENALI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-005
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: High-Grade Serous Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Keywords: Cyclin E1, CCNE1, Ovarian Cancer, Platinum Resistant, WEE1 inhibitor, DENALI, GOG-3066
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1a/1b (Arm completed enrollment); Part 2a-Arm 1 (Enrolling); Part 2a-Arm 2 (Enrolling); Part 2b (Arm not yet recruiting)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1a/1b (Completed Enrollment) (Experimental): Azenosertib 400mg administered on a 5 days on, 2 days off intermittent schedule.
  Interventions: Drug: azenosertib
- Part 2a: Arm 1 (Experimental): Azenosertib 400mg administered on a 5 days on, 2 days off intermittent schedule
  Interventions: Drug: azenosertib
- Part 2a: Arm 2 (Experimental): Azenosertib 300mg administered on a 5 days on, 2 days off intermittent schedule
  Interventions: Drug: azenosertib
- Part 2b (Experimental): Azenosertib at the dose selected in Part 2a administered on a 5 days on, 2 days off intermittent schedule
  Interventions: Drug: azenosertib

INTERVENTIONS:
Drug: azenosertib — Azenosertib (ZN-c3) will be administered orally.
  Other Names: ZN-c3

SUMMARY:
This is a multi-part Phase 2 study to evaluate the efficacy and safety of azenosertib (ZN-c3) in subjects with Platinum-Resistant, High-Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer. Part 2 of the study will be conducted in subjects whose tumors are Cyclin E1 positive as determined by central review using the Sponsor's investigational clinical trial assay.

DETAILED DESCRIPTION:
A Phase 2 study to evaluate the efficacy and safety of azenossertib (ZN-c3) in subjects with Platinum-Resistant, High-Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer. Azenosertib is a selective and orally bioavailable inhibitor of WEE1. By inhibiting WEE1, azenosertib enables cell cycle progression, despite high levels of DNA damage, thereby resulting in the accumulation of DNA damage leading to mitotic catastrophe and cancer cell death.

The study consists of two parts:

Part 1: All comers, no biomarker status required (completed enrollment)

Part 2: Cyclin E1 positive protein expression required

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. High-grade serous ovarian, fallopian tube or primary peritoneal cancer
3. Tumor testing (archival acceptable) confirms a positive Cyclin E1 protein status result determined by IHC using the Sponsor's investigational clinical trial assay
4. Prior therapy:

   1. Subjects must have platinum-resistant disease
   2. One to 3 prior lines or regimens are allowed (1 to 4 prior lines are permitted, if prior mirvetuximab)
   3. Prior bevacizumab treatment is required, if eligible per standard of care
   4. Prior PARP inhibitor treatment is required if BRCA 1/2 mutation or HRD, if eligible per standard of care
   5. Prior mirvetuximab treatment is required, if eligible per standard of care
5. Measurable disease per RECIST Version 1.1.
6. Adequate hematologic and organ function, as defined in protocol
7. ECOG 0-1

Exclusion Criteria:

1. Primary platinum-refractory disease
2. Any of the following treatment interventions within the specified time frame prior to C1D1:

   1. Major surgery within 28 days
   2. Hospitalization within 14 days
   3. Any chemotherapy or targeted tumor therapy within 21 days or 5 half-lives (whichever is shorter);
   4. Radiation therapy within 21 days;
   5. Autologous or allogeneic stem cell transplant within 3 months.
   6. Current use of any other investigational drug therapy <28 days or 5 half-lives (whichever is shorter).
   7. Inability to discontinue treatment prescription or non-prescription drugs, or to discontinue consumption of food and herbal supplements that are strong or moderate CYP3A inhibitors and inducers or P-gp inhibitors at least 14 days prior to C1D1.
3. Prior therapy with ZN-c3 or any other WEE1 inhibitor, ATR inhibitor, PKMYT1 inhibitor, or CHK1/2 inhibitor.
4. A serious illness or medical condition(s) including, but not limited to:

   1. Clinically or radiographically unstable brain metastases or leptomeningeal disease that requires immediate treatment. Subjects with asymptomatic brain metastases are eligible.
   2. Myocardial impairment resulting in heart failure (NYHA Class II-IV)
   3. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or may interfere with interpretation of study results
   4. Acute kidney injury requiring intervention or intravenous fluid in the last 14 days or presence of indwelling urinary catheter or percutaneous nephrostomy.
   5. Significant gastrointestinal abnormalities, including an inability to take oral medication, requirement for intravenous alimentation, active peptic ulcer, chronic diarrhea or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption.
   6. Active, uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal, or antiviral) must have completed such treatment and the infection must be considered controlled/resolved (and afebrile) by the Investigator for at least 7 days before C1D1
   7. Any evidence of bowel obstruction as determined by air/fluid levels on computed tomography (CT scan, recent hospitalization for small bowel obstruction within 3 months prior to C1D1, or recurrent paracentesis or thoracentesis within 6 weeks prior to C1D1.
5. Unresolved toxicity of Grade >1 attributed to any prior therapies (excluding Grade ≤2 neuropathy, alopecia, or skin pigmentation).
6. Pregnant or lactating female subject or female subject of childbearing potential who has a positive serum pregnancy test within 14 days prior to C1D1.
7. History of another malignancy in the previous 2 years, unless cured by surgery alone and continuously disease free. Exceptions include appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, or other malignancies with an expected curative outcome.
8. Subjects who are known to be immunocompromised or HIV-positive on highly active anti-retroviral therapy.
9. Subjects with known active hepatitis B or hepatitis C infection.
10. Individuals who are judged by the Investigator to be unsuitable as study subjects.
11. Subjects who had prior wide-field radiotherapy affecting ≥ 20% of the bone marrow.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) defined by RECIST v1.1 [Part 2] | Up to approximately 12 months from the enrollment of the last subject
  Participants who achieve partial response (PR) or complete response (CR) per RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) defined by RECIST v1.1 [Part 2] | Up to approximately 12 months from the enrollment of the last subject
  Time from the date of first documented response (CR or PR that is subsequently confirmed per RECIST v1.1) until the date of progressive disease (PD) or death.
Progression free survival (PFS) defined by RECIST v1.1 [Part 2] | Up to approximately 12 months from the enrollment of the last subject
  Time from the date of first dose until the date of PD or death.
Clinical Benefit Rate (CBR) defined by RECIST v1.1 [Part 2] | Up to approximately 12 months from the enrollment of the last subject
  The percentage of participants who have at least 1 confirmed response of CR or PR, or stable disease for at least 16 weeks before any evidence of progression.
CA-125 response by GCIG criteria [Part 2] | Up to approximately 12 months from the enrollment of the last subject
  The GCIG CA-125 response was defined as at least 50% reduction in CA-125 levels from baseline.
Number of Subjects experiencing treatment emergent adverse events (TEAEs) [Part 2] | Up to approximately 12 months from the enrollment of the last subject

CONTACTS AND LOCATIONS:
Locations (88):
- United States (44):
  - Site 0170-USA Mitchell Cancer Institute, Mobile, Alabama
  - Site 0143 - HonorHealth, Phoenix, Arizona
  - Site 0102 - University of Arizona Cancer Center, Tucson, Arizona
  - Site 0258 - UC San Diego Moores Cancer Center, La Jolla, California
  - Site 0287 - Ridley Tree Cancer Center, Santa Barbara, California
  - Site 0135 - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Site 0158 - Hartford HealthCare, Hartford, Connecticut
  - Site 0239 - Florida Cancer Specialists - East, Daytona Beach, Florida
  - Site 0173 - Mount Sinai Medical Center, Miami Beach, Florida
  - Site 0308 - Advent Health, Orlando, Florida
  - Site 0108 - Emory University Hospital, Atlanta, Georgia
  - Site 0236 - Memorial Health, Savannah, Georgia
  - Site 0324 - Illinois Cancer Specialists, Niles, Illinois
  - Site 0284 - Community Cancer Center North, Indianapolis, Indiana
  - Site 0217 - St Vincent Hospital and Health Care Centers, Indianapolis, Indiana
  - Site 0251 - Norton Cancer Institute, Louisville, Kentucky
  - Site 0146 - Maryland Oncology Hematology, PA, Rockville, Maryland
  - Site 0221 - Tufts Medical Center - PPDS, Boston, Massachusetts
  - Site 0104 - Dana Farber Cancer Institute, Boston, Massachusetts
  - Site 0307 - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Site 0263 - Baystate Medical Center, Springfield, Massachusetts
  - Site 0101 - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Site 0228 - Corewell Health Medical Group West, Grand Rapids, Michigan
  - Site 0288 - Minnesota Oncology Hematology - Maplewood, Maplewood, Minnesota
  - Site 0226 - CoxHealth, Springfield, Missouri
  - Site 0317 - Nebraska Methodist Hospital, Omaha, Nebraska
  - Site 0213 - Center of Hope, Reno, Nevada
  - Site 0231 - Northwell Health Cancer Institute, Manhasset, New York
  - Site 0126 - Wilmot Cancer Center, Rochester, New York
  - Site 0259 - Duke Cancer Center, Durham, North Carolina
  - Site 0147 - Trihealth Cancer Institute - Harold and Eugen, Cincinnati, Ohio
  - Site 0243 - Mark H Zangmeister Cancer Center, Columbus, Ohio
  - Site 0214-Ohio State University Comprehensive Cancer Center, Hilliard, Ohio
  - Site 0316 - Willamette Valley Cancer Institute/Oncology Associates of Oregon, Eugene, Oregon
  - Site 0232 - University of Pennsylvania, Philadelphia, Pennsylvania
  - Site 0178 - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Site 0277 - Alliance Cancer Specialist, PC, Wynnewood, Pennsylvania
  - Site 0132 - Avera Cancer Institute, Sioux Falls, South Dakota
  - Site 0103 - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Site 0234 - University of Texas Health, Memorial Hermann Hospital, Houston, Texas
  - Site 0203 - Texas Oncology, Tyler, Texas
  - Site 0295 - Virginia Oncology Associates, Chesapeake, Virginia
  - Site 0322 - Inova Schar Cancer Institute, Fairfax, Virginia
  - Site 0323 - Compass Oncology, Vancouver, Washington
- Australia (7):
  - Site 2715 - Icon Cancer Centre - Chermside, Chermside, Queensland
  - Site 2707 - Mater Brisbane, South Brisbane, Queensland
  - Site 2709 - Cancer Research SA, Adelaide, South Australia
  - Site 2702 - Burnside War Memorial Hospital - The Brian Fricker Oncology Centre, Toorak Gardens, South Australia
  - Site 2716 - Epworth Healthcare Freemasons, East Melbourne, Victoria
  - Site 2701 - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Site 2717 - St John of God Hospital Subiaco, Subiaco, Western Australia
- Belgium (3):
  - Site 3102 - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Site 3101 - AZORG - Aalst, Aalst, Oost-Vlaanderen
  - Site 3105 - UZ Leuven, Leuven, Vlaams Brabant
- France (13):
  - Site 3616 - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - Site 3611 - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg, Bas-Rhin
  - Site 3601 - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Site 3613 - CHRU Besancon - Hopital Jean Minjoz, Besançon, Doubs
  - Site 3617 - CHU de Brest - Hôpital La Cavale Blanche, Brest, Finistere
  - Site 3603 - Institut Claudius Regaud, Toulouse, Haute-Garonne
  - Site 3602 - Centre Oscar Lambret, Lille, Nord
  - Site 3615 - Hôpital Cochin Port-Royal AP-HP, Paris, Paris
  - Site 3614 - Institut de Cancerologie de l'oust, Saint-Herblain, Pays de la Loire Region
  - Site 3608 - Hospices Civils de Lyon - Hôpital Lyon Sud, Pierre-Bénite, Rhône
  - Site 3619 - Centre Léon Bérard, Lyon
  - Site 3620 - CHU de Strasbourg - Hopital de Hautepierre, Strasbourg
  - Site 3604 - Institut Gustave Roussy, Villejuif
- Italy (8):
  - Site 3302 - Istituto Nazionale Tumori IRCCS Fondazione Giovanni Pascale, Napoli, Campania
  - Site 3308 - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Site 3312 - Centro di Riferimento Oncologico, Aviano, Friuli Venezia Giulia
  - Site 3304 - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Site 3305 - Istituto Europeo di Oncologia, Milan, Lombardy
  - Site 3307 - Ospedale San Raffaele S.r.l., Milan, Milano
  - Site 3311 - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - Site 3303 - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi-Via Massarenti, Bologna
- Poland (5):
  - Site 2414 - Med-Polonia Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Site 2405 - Centrum Badan Klinicznych JCI, Krakow, Lesser Poland Voivodeship
  - Site 2404 - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Site 2419 - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Site 2421 - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
- South Korea (3):
  - Site 2909 - Severance Hospital Yonsei University Health System, Seoul
  - Site 2906 - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Site 2907 - Samsung Medical Center, Seoul
- Spain (5):
  - Site 3511 - Instituto de Investigacion Oncologica Vall d'Hebron, Barcelona, Barcelona
  - Site 3517 - Clinica Universidad de Navarra, Madrid, Madrid
  - Site 3516 - Hospital Universitario Virgen de La Arrixaca, Murcia, Murcia
  - Site 3501 - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Site 3502 - Hospital Universitario La Paz, Madrid